CLINICAL TRIAL: NCT04136236
Title: Automatic Diagnosis of Early Esophageal Squamous Neoplasia Using Probe-based Confocal Laser Endomicroscopy With Artificial Intelligence
Brief Title: Automatic Diagnosis of Early Esophageal Squamous Neoplasia Using pCLE With AI
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of QiLu Hospital, Shandong University
Other Study IDs: 2019SDU-QILU-66
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Neoplasms; Artificial Intelligence; Confocal Laser Endomicroscopy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — When suspected lesion is found using white light endoscopy , endoscopist will observe this lesion using pCLE and then take biopsy for histology examination.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- esophageal mucosal lesions observed by pCLE: pCLE is used to distinguish the suspected lesions detected by white light endoscopy or IEE.
  Interventions: Diagnostic Test: The diagnosis of Artificial Intelligence and endoscopist

INTERVENTIONS:
Diagnostic Test: The diagnosis of Artificial Intelligence and endoscopist — Suspected esophageal mucosal lesion is observed using pCLE, endoscopist and AI will make a diagnosis independently. In addition, the endoscopist can not see the diagnosis of AI. After a washout period, nonexpert endoscopists take the second assessment with AI assistance.

SUMMARY:
Detection and differentiation of esophageal squamous neoplasia (ESN) are of value in improving patient outcomes. Probe-based confocal laser endomicroscopy (pCLE) can diagnose ESN accurately.However this requires much experience, which limits the application of pCLE. The investigators designed a computer-aided diagnosis program using deep neural network to make diagnosis automatically in pCLE examination and contrast its performance with endoscopists.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80;
* agree to give written informed consent；

Exclusion Criteria:

* advanced esophageal squamous cell carcinoma or esophageal stenosis;
* having no suspicious lesion of ESN found by WLE and IEE
* known allergy to fluorescein sodium;
* having coagulopathy or impaired renal function;
* being pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who receive the upper gastrointestinal tract pCLE examination and screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
The diagnosis efficiency of Artificial Intelligence | 3 years
  The primary outcome is to test the diagnostic accuracy, sensitivity, specificity, PPV, NPV of the Artificial Intelligence for diagnosing esophageal mucosal disease on real-time pCLE examination.

SECONDARY OUTCOMES:
Contrast the diagnosis efficiency of Artificial Intelligence with endoscopists | 1 month
  The secondary outcome is to compare the diagnosis efficiency (including diagnostic accuracy, sensitivity, specificity, PPV, NPV for diagnosing esophageal mucosal disease on real-time pCLE examination) between Artificial Intelligence and endoscopists.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China